CLINICAL TRIAL: NCT02644174
Title: The Impact of Bariatric Surgery Induced Weight Loss on Lung Function in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Stafler, Dr, Rabin Medical Center
Other Study IDs: 0126-16-RMC
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Obesity; Lung function test; Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bariatric Surgery

SUMMARY:
In this prospective study we will evaluate the changes in respiratory physiology occurring in morbidly obese adolescents following bariatric surgery at Schneider Children's Medical Center of Israel (SCMCI).

DETAILED DESCRIPTION:
Morbid obesity leads to restrictive as well as obstructive ventilatory defects via mechanisms that include mechanical, as well as inflammatory factors. We hypothesise that multiple breath nitrogen washout will be more sensitive to changes in small airway function than conventional lung function testing.

We will invite adolescents with morbid obesity, scheduled to undergo bariatric surgery at SCMCI during 2016-2018, for pulmonary function testing, including spirometry, plethysmography, nitrogen multiple breath washout, lung transfer factor and 6 minute walk. These tests will be conducted prior to the operation as well as during follow-up appointments at 3, 6 and 12 months. We will also evaluate oxidative stress using highly sensitive C-reactive protein as surrogate marker.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with morbid obesity who will undergo bariatric surgery at the paediatric surgery ward of Schneider Children's Medical Center during 2016-2018

Exclusion Criteria:

* Adolescents with background diseases which might influence their ability to conduct pulmonary function tests (for example, patients with neurological disorders)

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with morbid obesity who will undergo bariatric surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Lung Clearance Index | 3 months post op

SECONDARY OUTCOMES:
Change from Baseline High sensitivity C reactive protein | 3 months post op

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed journal

REFERENCES:
- [Background] Li AM, Chan D, Wong E, Yin J, Nelson EA, Fok TF. The effects of obesity on pulmonary function. Arch Dis Child. 2003 Apr;88(4):361-3. doi: 10.1136/adc.88.4.361. PMID 12651773
- [Background] Lazarus R, Colditz G, Berkey CS, Speizer FE. Effects of body fat on ventilatory function in children and adolescents: cross-sectional findings from a random population sample of school children. Pediatr Pulmonol. 1997 Sep;24(3):187-94. doi: 10.1002/(sici)1099-0496(199709)24:33.0.co;2-k. PMID 9330415
- [Background] Kelleher DC, Merrill CT, Cottrell LT, Nadler EP, Burd RS. Recent national trends in the use of adolescent inpatient bariatric surgery: 2000 through 2009. JAMA Pediatr. 2013 Feb;167(2):126-32. doi: 10.1001/2013.jamapediatrics.286. PMID 23247297
- [Background] Kalra M, Inge T, Garcia V, Daniels S, Lawson L, Curti R, Cohen A, Amin R. Obstructive sleep apnea in extremely overweight adolescents undergoing bariatric surgery. Obes Res. 2005 Jul;13(7):1175-9. doi: 10.1038/oby.2005.139. PMID 16076986
- [Background] Abu-Abeid S, Gavert N, Klausner JM, Szold A. Bariatric surgery in adolescence. J Pediatr Surg. 2003 Sep;38(9):1379-82. doi: 10.1016/s0022-3468(03)00400-7. PMID 14523824
- [Background] Weiner P, Waizman J, Weiner M, Rabner M, Magadle R, Zamir D. Influence of excessive weight loss after gastroplasty for morbid obesity on respiratory muscle performance. Thorax. 1998 Jan;53(1):39-42. doi: 10.1136/thx.53.1.39. PMID 9577520
- [Background] Davila-Cervantes A, Dominguez-Cherit G, Borunda D, Gamino R, Vargas-Vorackova F, Gonzalez-Barranco J, Herrera MF. Impact of surgically-induced weight loss on respiratory function: a prospective analysis. Obes Surg. 2004 Nov-Dec;14(10):1389-92. doi: 10.1381/0960892042583996. PMID 15603656
- [Background] Santana AN, Souza R, Martins AP, Macedo F, Rascovski A, Salge JM. The effect of massive weight loss on pulmonary function of morbid obese patients. Respir Med. 2006 Jun;100(6):1100-4. doi: 10.1016/j.rmed.2005.09.021. Epub 2005 Oct 21. PMID 16243500
- [Background] Nguyen NT, Hinojosa MW, Smith BR, Gray J, Varela E. Improvement of restrictive and obstructive pulmonary mechanics following laparoscopic bariatric surgery. Surg Endosc. 2009 Apr;23(4):808-12. doi: 10.1007/s00464-008-0084-9. Epub 2008 Sep 20. PMID 18806943
- [Background] Sahebjami H, Gartside PS. Pulmonary function in obese subjects with a normal FEV1/FVC ratio. Chest. 1996 Dec;110(6):1425-9. doi: 10.1378/chest.110.6.1425. PMID 8989055
- [Background] Rubinstein I, Zamel N, DuBarry L, Hoffstein V. Airflow limitation in morbidly obese, nonsmoking men. Ann Intern Med. 1990 Jun 1;112(11):828-32. doi: 10.7326/0003-4819-112-11-828. PMID 2378649
- [Background] Hakala K, Mustajoki P, Aittomaki J, Sovijarvi AR. Effect of weight loss and body position on pulmonary function and gas exchange abnormalities in morbid obesity. Int J Obes Relat Metab Disord. 1995 May;19(5):343-6. PMID 7647827
- [Background] Thomas PS, Cowen ER, Hulands G, Milledge JS. Respiratory function in the morbidly obese before and after weight loss. Thorax. 1989 May;44(5):382-6. doi: 10.1136/thx.44.5.382. PMID 2503905
- [Background] Vaughan RW, Cork RC, Hollander D. The effect of massive weight loss on arterial oxygenation and pulmonary function tests. Anesthesiology. 1981 Apr;54(4):325-8. doi: 10.1097/00000542-198104000-00013. PMID 7212333
- [Background] Sugerman HJ, Baron PL, Fairman RP, Evans CR, Vetrovec GW. Hemodynamic dysfunction in obesity hypoventilation syndrome and the effects of treatment with surgically induced weight loss. Ann Surg. 1988 May;207(5):604-13. doi: 10.1097/00000658-198805000-00015. PMID 3377570
- [Background] Boone KA, Cullen JJ, Mason EE, Scott DH, Doherty C, Maher JW. Impact of Vertical Banded Gastroplasty on Respiratory Insufficiency of Severe Obesity. Obes Surg. 1996 Dec;6(6):454-458. doi: 10.1381/096089296765556322. PMID 10729891
- [Background] Scheuller M, Weider D. Bariatric surgery for treatment of sleep apnea syndrome in 15 morbidly obese patients: long-term results. Otolaryngol Head Neck Surg. 2001 Oct;125(4):299-302. doi: 10.1067/mhn.2001.119139. PMID 11593162
- [Background] Dixon JB, Schachter LM, O'Brien PE. Polysomnography before and after weight loss in obese patients with severe sleep apnea. Int J Obes (Lond). 2005 Sep;29(9):1048-54. doi: 10.1038/sj.ijo.0802960. PMID 15852048
- [Background] Aaron SD, Fergusson D, Dent R, Chen Y, Vandemheen KL, Dales RE. Effect of weight reduction on respiratory function and airway reactivity in obese women. Chest. 2004 Jun;125(6):2046-52. doi: 10.1378/chest.125.6.2046. PMID 15189920